CLINICAL TRIAL: NCT00701129
Title: An Exploratory Study of the Safety and Efficacy of Prophylactic Immunomodulatory Treatment in Myozyme®-Naive, CRIM(-) Patients With Infantile-onset Pompe Disease
Brief Title: An Exploratory Study of the Safety and Efficacy of Prophylactic Immunomodulatory Treatment in Myozyme-naive Cross-Reacting Immunologic Material (CRIM[-]) Patients With Infantile-Onset Pompe Disease
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Genzyme, a Sanofi Company (Industry)
Responsible Party: Sponsor
Organization: Sanofi (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AGLU03807; MSC12862 (Other: Sanofi)
Record Dates: First submitted 2008-06-17; First posted 2008-06-19 (Estimated); Results first posted 2014-05-13 (Estimated); Last update posted 2014-05-13 (Estimated); Status verified 2014-04

CONDITIONS: Pompe Disease; Glycogen Storage Disease Type II
Keywords: Glycogenesis 2; Acid; Maltase; Deficiency
MeSH Terms: conditions — Glycogen Storage Disease Type II; Heartburn | interventions — GAA protein, human; Methotrexate; Rituximab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Alglucosidase Alfa (Experimental): Alglucosidase alfa (Myozyme®) 20 milligrams per kilogram (mg/kg) intravenous (IV) infusion every other week (qow) (or optionally 20 mg/kg IV infusion every week [qw]) beginning from Day 0 to a minimum of 18 months or if the patient was less than (<) 6 months of age at the time of enrollment, until the patient was 2 years of age, along with methotrexate 0.4 mg/kg subcutaneously for 3 consecutive days qow beginning from Day 0 to Week 6 (9 doses) and rituximab 375 milligrams per square meter (mg/m^2) (or 12.5 mg/kg for patients with body surface area less than or equal to 0.5 m^2) IV infusion qw beginning from Day -1 to Week 4 (4 doses) as per local prescribing information. An additional 4-week cycle of rituximab (up to 4 additional doses) and 6-week cycle of methotrexate (up to 9 additional doses) may have been administered within the first 6 months of the study as per local prescribing information.
  Interventions: Biological: Alglucosidase Alfa; Drug: Methotrexate; Drug: Rituximab

INTERVENTIONS:
Biological: Alglucosidase Alfa — Administered as IV infusion.
  Other Names: Myozyme®
Drug: Methotrexate — Administered subcutaneously.
Drug: Rituximab — Administered as IV infusion.

SUMMARY:
The purpose of this study was to evaluate the efficacy, clinical benefits and safety of a prophylactic immunomodulatory regimen given prior to first treatment with alglucosidase alfa (Myozyme®) in patients with infantile-onset Pompe disease.

The objectives were to assess the efficacy of a prophylactic immunomodulatory regimen given prior to first treatment with alglucosidase alfa, as assessed by anti-recombinant human acid alpha-glucosidase (anti-rhGAA) antibody titers, and antibodies that inhibit the activity and/or uptake of alglucosidase alfa; to evaluate the clinical benefit as measured by overall survival, ventilator-free survival, left ventricular mass index (LVMI), gross motor function and development, disability index and the incidence of adverse events (AEs), serious adverse events (SAEs), and clinical laboratory abnormalities.

ELIGIBILITY:
Inclusion Criteria:

* The patient's legal guardian(s) must have provided written informed consent prior to any study-related procedures being performed
* The patient must have had a clinical diagnosis of Pompe disease as defined by documented acid alpha-glucosidase (GAA) deficiency (deficient endogenous GAA activity) in skin fibroblasts, muscle, or blood, or 2 GAA mutations. Consent was also sought from the biological parent(s) for parental GAA mutational analysis, but was not a requirement for study eligibility
* The patient must have not received Myozyme® or any rhGAA therapies prior to enrollment in the study
* The patient must be CRIM negative via Western Blot analysis performed on skin fibroblasts or via 2 known CRIM negative mutations (in which case CRIM status was to be confirmed by Western Blot analysis after enrollment)
* The patient's legal guardian(s) must have the ability to comply with the clinical protocol

Exclusion Criteria:

* The patient had any medical condition that, in the opinion of the Investigator, could be exacerbated/precipitated by or interfere with the study regimen or assessments; such conditions may include but were not limited to human immunodeficiency virus, cancer, Hepatitis B, Hepatitis C, Cytomegalovirus, Herpes Simplex, John Cunningham (JC) virus, Parvovirus, or Epstein Barr virus or tuberculosis
* The patient had used any investigational product within 30 days prior to study enrollment
* The patient had or was required to have any live vaccination within 1 month prior to enrollment

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2009-10; Primary Completion 2013-03 (Actual); Study Completion 2013-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Genzyme Coorporation
Locations (2):
- United States (2):
  - Kosair Children's Hospital, Louisville, Kentucky
  - Duke University Medical Center, Durham, North Carolina

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted at 2 centers in the United States of America between October 01, 2009 and March 27, 2013.
Period: Overall Study
Arm/Group | Alglucosidase Alfa
Started | 4
Full Analysis Set (FAS) | 4 (All enrolled patients who signed informed consent, received at least 1 dose of alglucosidase alfa.)
Completed | 2
Not Completed | 2
Not completed — Death | 2

BASELINE CHARACTERISTICS:
Population: Safety population included all patients who received at least one dose of alglucosidase alfa.
Groups:
- Alglucosidase Alfa: Alglucosidase alfa (Myozyme®) 20 mg/kg IV infusion qow (or optionally 20 mg/kg IV infusion every week [qw]) beginning from Day 0 to a minimum of 18 months or if the patient was <6 months of age at the time of enrollment, until the patient was 2 years of age, along with methotrexate 0.4 mg/kg subcutaneously for 3 consecutive days qow beginning from Day 0 to Week 6 (9 doses) and rituximab 375 mg/m^2 (or 12.5 mg/kg for patients with body surface area less than or equal to 0.5 m^2) IV infusion qw beginning from Day -1 to Week 4 (4 doses) as per local prescribing information. An additional 4-week cycle of rituximab (up to 4 additional doses) and 6-week cycle of methotrexate (up to 9 additional doses) may have been administered within the first 6 months of the study as per local prescribing information.
Arm/Group | Alglucosidase Alfa
Number analyzed (Participants) | 4
Age, Customized [Number; unit: participants]
  Less Than or Equal to (=<) 6 Months | 2
  Greater Than (>) 6 Months | 2
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3
  Male | 1
Race/Ethnicity, Customized [Number; unit: participants]
  Race: Black | 2
  Race: White | 1
  Race: White, Black | 1
  Ethnicity: Hispanic | 2
  Ethnicity: Non Hispanic | 2
Number of Patients With Anti-Recombinant Human Acid Alfa-glucosidase (Anti-rhGAA) Immunoglobulin G [Number; unit: participants] — As all patients were treatment naïve, it was expected that no patient would be Anti-rhGAA immunoglobulin G (IgG) antibody positive at baseline.
  participants
    Negative | 4
    Positive | 0
Number of Patients With Normal/Abnormal Left Ventricular Mass (LVM) Z-Score and LVM Index [Number; unit: participants] — LVM Z-Score and LVM Index were assessed by echocardiography (ECHO). LVM Z-Score: an indicator of degree of standard deviations from mean in a normal distribution. Negative values indicate a smaller LVM than mean and values higher than 0 indicate a larger LVM than mean. Normal range is -2 to 2; values <-2 or >2 indicate abnormal score. LVM index: an index value derived by normalizing LVM by body surface area. LVM index provides evidence of cardiomyopathy. LVM index values <65 gram per square meter (g/m^2) were considered as normal and LVM index values >=65 g/m^2 were considered as abnormal.
  participants
    LVM Z-score: Normal | 0
    LVM Z-score: Abnormal | 4
    LVM index: Normal | 0
    LVM index: Abnormal | 4
Number of Patients With Ventilator Use [Number; unit: participants]
  Yes | 3
  No | 1
Gross Motor Disability Assessed by Gross Motor Function Measure-88 (GMFM-88) [Median (Full Range); unit: percentage of maximum total score] — GMFM-88:an 88-item measure to detect gross motor function; consists of 5 categories: lying and rolling; sitting; crawling and kneeling; standing; walking, running and jumping. Each item is scored on a 4-point Likert scale(0=cannot do; 1=initiates [<10% of the task]; 2=partially completes [10% to <100% of the task]; 3=task completion). Score for each dimension is expressed as a percentage of maximum score for that dimension. Total score=sum of percentage scores for each dimension divided by number of dimensions. Total score range: 0% to 100%, where higher scores indicate better motor functions.
  percentage of maximum total score | 5.10 [0.39 to 7.49]
Motor Development Status Assessed by Alberta Infantile Motor Scale (AIMS) [Median (Full Range); unit: months] — AIMS:58-item in 4 subscales: prone; supine; sitting; and standing. Each item is scored as observed/not observed. Item in observed range create a motor window. Subscale scores are calculated by giving child 1 point for observed items within motor window in addition to being given 1 point for all less mature items before motor window. AIMS total score=sum of scores for 58 items, range: 0-58,higher score=more mature motor development. Score was then compared with age-equivalent peers from normative sample and equivalence level age (in months) is reported. Here, number of patients analyzed = 3.
  months | 0 [0 to 1.37]
Disability Index Assessed by the Pompe Pediatric Evaluation of Disability Inventory (Pompe PEDI) [Median (Full Range); unit: units on a scale] — It consists of all items of original PEDI (197 functional skill items in 3 domains:self-care;mobility;social function) and additional items in functional skills,mobility,self-care domains to reflect functional skills for children with Pompe. Each domain consists of 2 subdomains: functional skill performance, caregiver assistance scale. Norm-based scoring was developed for additional items, and scoring for PEDI have been adjusted to reflect additional normative data collected for Pompe PEDI. Total score range for each domain (mean of subdomains) and subdomain=0-100;higher score=high capability.
  units on a scale
    Functional Skills: Mobility Score (n=4) | 4.5 [0 to 18.4]
    Functional Skills: Self-Care Score (n=4) | 14.4 [4.9 to 16.1]
    Functional Skills: Social Function Score (n=1) | 10.5 [10.5 to 10.5]
    Caregiver Assistance: Mobility Score (n=2) | 0 [0 to 0]
    Caregiver Assistance: Self-Care Score (n=2) | 0 [0 to 0]
    Caregiver Assistance: Social Function Score (n=2) | 0 [0 to 0]

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Number of Patients With Anti-Recombinant Human Acid Alfa-glucosidase (Anti-rhGAA) Immunoglobulin G (IgG) Antibody at End of Study
Description: Serum samples from patients were analyzed for the presence of anti-rhGAA IgG antibodies. End of study (EOS) refers to the last post baseline observation during study period (up to Week 79).
Time Frame: Baseline, End of Study (up to Week 79 or early termination)
Population: FAS population included all enrolled patients who signed informed consent and received at least 1 dose of alglucosidase alfa.
Measure: Number; unit: participants
Arm/Group | Alglucosidase Alfa
Number analyzed (Participants) | 4
participants
  Baseline - Negative; EOS - Positive | 2
  Baseline - Negative; EOS - Negative | 2

2. Primary Outcome: Number of Patients With Recombinant Human Acid Alfa-glucosidase (rhGAA) Inhibitory Antibody at End of Study
Description: Patients with positive anti-rhGAA IgG antibody were assessed for the presence of inhibitory antibodies (inhibition of enzyme activity and inhibition of enzyme uptake). Enzyme-linked immunosorbent assay (ELISA) was used to measure inhibition of rhGAA enzymatic activity in vitro and a cell-based assay was used to measure the inhibition of the uptake of rhGAA in normal fibroblast cells by flow cytometry.
Time Frame: End of study (up to Week 79)
Population: FAS population included all enrolled patients who signed informed consent and received at least 1 dose of alglucosidase alfa. Here, number of patients analyzed = patients with positive anti-rhGAA IgG antibody.
Measure: Number; unit: participants
Arm/Group | Alglucosidase Alfa
Number analyzed (Participants) | 2
participants
  Inhibition of Enzyme Activity | 0
  Inhibition of Enzyme Uptake | 0

3. Primary Outcome: Number of Patients Who Survived at End of Study
Time Frame: Baseline up to End of study (Week 79)
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | Alglucosidase Alfa
Number analyzed (Participants) | 4
participants | 2

4. Primary Outcome: Number of Patients With Normal/Abnormal Left Ventricular Mass (LVM) Z-Score and LVM Index at End of Study
Description: LVM Z-score and LVM index were assessed by ECHO. LVM Z-Score provides an indicator of degree of standard deviations from the mean in a normal distribution. Negative values indicate a smaller LVM than mean and values higher than 0 indicate a larger LVM than the mean. The normal range for LVM Z-Score is -2 to 2. Values <-2 or >2 indicate abnormal LVM Z-Score. LVM index is an index value derived by normalizing LVM by body surface area. LVM index provides evidence of cardiomyopathy. LVM index values <65 gram per meter^2 (g/m^2) were considered as normal and LVM index values >=65 g/m^2 were considered as abnormal. End of study refers to the last post baseline observation during study period (up to Week 79).
Time Frame: End of study (up to Week 79 or early termination)
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | Alglucosidase Alfa
Number analyzed (Participants) | 4
participants
  LVM Z-score: Normal | 3
  LVM Z-score: Abnormal | 1
  LVM index: Normal | 2
  LVM index: Abnormal | 2

5. Primary Outcome: Number of Patients With Ventilator Use at End of Study
Description: Number of patients who had ventilator support at end of study was reported. End of study refers to the last post baseline observation during study period (up to Week 79).
Time Frame: End of study (up to Week 79 or early termination)
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | Alglucosidase Alfa
Number analyzed (Participants) | 4
participants
  Yes | 3
  No | 1

6. Primary Outcome: Gross Motor Disability Assessed by Gross Motor Function Measure-88 (GMFM-88) at End of Study
Description: GMFM-88 is an 88-item measure to detect gross motor function. It consists of 5 categories: lying and rolling; sitting; crawling and kneeling; standing; walking, running and jumping. Each item is scored on a 4-point Likert scale (0 = cannot do; 1 = initiates [<10% of the task]; 2 = partially completes [10% to <100% of the task]; 3 = task completion). The score for each dimension is expressed as a percentage of the maximum score for that dimension. Total score is obtained by adding the percentage scores for each dimension and dividing the sum by the total number of dimensions. Total score ranges from 0% to 100%, where higher scores indicate better motor functions. A total score of <7.5% demonstrates gross motor disability. End of study refers to the last post baseline observation during study period (up to Week 79).
Time Frame: End of study (up to Week 79 or early termination)
Population: FAS population included all enrolled patients who signed informed consent and received at least 1 dose of alglucosidase alfa. Here, numbers of patients analyzed = patients with end of study GMFM-88 assessment.
Measure: Median (Full Range); unit: percentage of maximum total score
Arm/Group | Alglucosidase Alfa
Number analyzed (Participants) | 3
percentage of maximum total score | 8.24 [6.76 to 89.8]

7. Primary Outcome: Motor Development Status Assessed by Alberta Infantile Motor Scale (AIMS) at End of Study
Description: AIMS is a 58-item reliable and valid measure of motor development for infants at risk for motor delay. It assesses infant movement in 4 positions (subscales): prone (reciprocal crawling); supine (moving hands to feet); sitting (sitting with arm support); and standing (pulls to stand). For each subscale, items were scored as "observed" or "not observed". Item in the observed range create a motor window. When scoring, subscale scores are calculated by giving the child credit (1 point) for observed items within the motor window in addition to being given credit (1 point) for all of the less mature items before motor window. AIMS total score was calculated by summing the scores for 58 items and ranged from 0 to 58, with higher score indicating more mature motor development. Score was then compared with age-equivalent peers from normative sample and equivalence level age (in months) is reported. End of study refers to the last post baseline observation during study period (up to Week 79).
Time Frame: End of study (up to Week 79 or early termination)
Population: FAS population included all enrolled patients who signed informed consent and received at least 1 dose of alglucosidase alfa. Here, numbers of patients analyzed = patients with end of study AIMS assessment.
Measure: Median (Full Range); unit: months
Arm/Group | Alglucosidase Alfa
Number analyzed (Participants) | 3
months | 1.09 [1.0 to 14.5]

8. Primary Outcome: Disability Index Assessed by the Pompe Pediatric Evaluation of Disability Inventory (Pompe PEDI) at End of Study
Description: The Pompe PEDI is a disease specific version of the PEDI that was developed to assess functional capabilities and performance in children with Pompe disease from 2 months through adolescence. It consists of all items of the original PEDI (197 functional skill items in 3 domains: self-care; mobility; and social function) and additional items in the functional skills, mobility, and self-care domains to reflect clinically relevant functional skills for children with Pompe disease. Each domain consisted of 2 subdomains: functional skill performance and caregiver assistance scale. Norm-based scoring was developed for these additional items, and scoring algorithms for the PEDI have been adjusted to reflect additional normative data collected for the Pompe PEDI. Total score range for each domain (mean of subdomains) and subdomain ranges from 0 to 100, where higher score indicates high capability. End of study refers to the last post baseline observation during study period (up to Week 79).
Time Frame: End of study (up to Week 79 or early termination)
Population: FAS population included all enrolled patients who signed informed consent and received at least 1 dose of alglucosidase alfa. Here, number of patient analyzed = number of patients with end of study Pompe PEDI assessment and n = number of patients with end of study assessment of specified category.
Measure: Median (Full Range); unit: units on a scale
Arm/Group | Alglucosidase Alfa
Number analyzed (Participants) | 3
units on a scale
  Functional Skills: Mobility Score (n=3) | 25.1 [23.2 to 56]
  Functional Skills: Self-Care Score (n=3) | 39.3 [37 to 55.2]
  Functional Skills: Social Function Score (n=3) | 46.2 [40.4 to 46.8]
  Caregiver Assistance: Mobility Score (n=3) | 20.3 [20.3 to 31.9]
  Caregiver Assistance: Self-Care Score (n=2) | 28.7 [20.1 to 37.2]
  Caregiver Assistance: Social Function Score (n=3) | 48.5 [20.4 to 53.1]

ADVERSE EVENTS:
Time Frame: First dose of study drug up to end of study (up to Week 79)
Description: In the event a single participant has experienced both serious and non-serious form of the same adverse event (AE), individual has been included in numerator of both AE tables. Analysis was performed on the safety population: all patients who received at least 1 dose of alglucosidase alfa. AEs are listed independent of relationship to treatment.
Arm/Group | Alglucosidase Alfa
Serious Adverse Events (participants affected / at risk) | 3/4
Other Adverse Events (participants affected / at risk) | 4/4
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Alglucosidase Alfa (N=4)
Arrhythmia (Cardiac disorders) | 1
Bradycardia (Cardiac disorders) | 1
Cardiac arrest (Cardiac disorders) | 1
Cardiopulmonary failure (Cardiac disorders) | 1
Tympanic membrane disorder (Ear and labyrinth disorders) | 1
Disease progression (General disorders) | 1
Pyrexia (General disorders) | 2
Clostridium difficile colitis (Infections and infestations) | 1
Pneumonia (Infections and infestations) | 1
Serratia sepsis (Infections and infestations) | 1
Tracheitis (Infections and infestations) | 1
Feeding tube complication (Injury, poisoning and procedural complications) | 1
Torus fracture (Injury, poisoning and procedural complications) | 1
Pulse absent (Investigations) | 1
Fluid imbalance (Metabolism and nutrition disorders) | 1
Muscle contracture (Musculoskeletal and connective tissue disorders) | 1
Apnoea (Respiratory, thoracic and mediastinal disorders) | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1
Laryngeal stenosis (Respiratory, thoracic and mediastinal disorders) | 1
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 2
Vena cava thrombosis (Vascular disorders) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Alglucosidase Alfa (N=4)
Anaemia (Blood and lymphatic system disorders) | 2
Lymphadenopathy (Blood and lymphatic system disorders) | 1
Neutropenia (Blood and lymphatic system disorders) | 1
Bradycardia (Cardiac disorders) | 2
Cyanosis (Cardiac disorders) | 1
Extrasystoles (Cardiac disorders) | 1
Tachycardia (Cardiac disorders) | 2
Tympanic membrane disorder (Ear and labyrinth disorders) | 2
Conjunctivitis (Eye disorders) | 1
Eyelid ptosis (Eye disorders) | 1
Periorbital oedema (Eye disorders) | 1
Anal sphincter atony (Gastrointestinal disorders) | 1
Anorectal disorder (Gastrointestinal disorders) | 1
Constipation (Gastrointestinal disorders) | 2
Diarrhoea (Gastrointestinal disorders) | 3
Duodenogastric reflux (Gastrointestinal disorders) | 1
Flatulence (Gastrointestinal disorders) | 1
Gastritis (Gastrointestinal disorders) | 1
Haematemesis (Gastrointestinal disorders) | 1
Haematochezia (Gastrointestinal disorders) | 1
Retching (Gastrointestinal disorders) | 1
Teething (Gastrointestinal disorders) | 1
Vomiting (Gastrointestinal disorders) | 3
Catheter site discharge (General disorders) | 1
Catheter site erosion (General disorders) | 1
Catheter site erythema (General disorders) | 2
Catheter site pruritus (General disorders) | 1
Catheter site rash (General disorders) | 2
Catheter site related reaction (General disorders) | 1
Device dislocation (General disorders) | 1
Device occlusion (General disorders) | 3
Face oedema (General disorders) | 1
Fatigue (General disorders) | 1
Intentional medical device removal by patient (General disorders) | 2
Medical device complication (General disorders) | 1
Oedema peripheral (General disorders) | 2
Pyrexia (General disorders) | 4
Body tinea (Infections and infestations) | 1
Candidiasis (Infections and infestations) | 1
Catheter site cellulitis (Infections and infestations) | 1
Clostridium difficile colitis (Infections and infestations) | 1
Gastroenteritis (Infections and infestations) | 1
Impetigo (Infections and infestations) | 1
Oral candidiasis (Infections and infestations) | 1
Otitis media (Infections and infestations) | 1
Otitis media acute (Infections and infestations) | 1
Sepsis (Infections and infestations) | 1
Serratia infection (Infections and infestations) | 1
Tracheitis (Infections and infestations) | 2
Urinary tract infection enterococcal (Infections and infestations) | 1
Viral infection (Infections and infestations) | 1
Burns second degree (Injury, poisoning and procedural complications) | 1
Laceration (Injury, poisoning and procedural complications) | 1
Lip injury (Injury, poisoning and procedural complications) | 1
Medication error (Injury, poisoning and procedural complications) | 1
Overdose (Injury, poisoning and procedural complications) | 1
Procedural pain (Injury, poisoning and procedural complications) | 2
Procedural site reaction (Injury, poisoning and procedural complications) | 1
Spinal compression fracture (Injury, poisoning and procedural complications) | 1
Torus fracture (Injury, poisoning and procedural complications) | 1
Alanine aminotransferase increased (Investigations) | 2
Antibiotic resistant Staphylococcus test positive (Investigations) | 1
Aspartate aminotransferase increased (Investigations) | 2
Band neutrophil percentage increased (Investigations) | 1
Blood chloride decreased (Investigations) | 1
Blood creatine phosphokinase MB increased (Investigations) | 2
Blood creatine phosphokinase increased (Investigations) | 1
Blood culture positive (Investigations) | 1
Blood immunoglobulin G increased (Investigations) | 2
Blood iron decreased (Investigations) | 1
Blood lactate dehydrogenase increased (Investigations) | 1
Blood potassium decreased (Investigations) | 1
Blood potassium increased (Investigations) | 1
Blood pressure increased (Investigations) | 1
Blood sodium decreased (Investigations) | 1
Body temperature increased (Investigations) | 1
Clostridium test positive (Investigations) | 1
Eosinophil percentage increased (Investigations) | 1
Heart rate decreased (Investigations) | 1
Heart rate irregular (Investigations) | 1
Lymphocyte percentage decreased (Investigations) | 2
Moraxella test positive (Investigations) | 1
Neutrophil count decreased (Investigations) | 1
Neutrophil percentage increased (Investigations) | 1
Occult blood positive (Investigations) | 2
Oxygen saturation decreased (Investigations) | 2
Protein total decreased (Investigations) | 1
Respiratory rate decreased (Investigations) | 1
Respiratory rate increased (Investigations) | 1
Reticulocyte percentage increased (Investigations) | 1
Specific gravity urine increased (Investigations) | 1
Urinary hexose tetrasaccharide increased (Investigations) | 1
Urine output decreased (Investigations) | 1
Weight decreased (Investigations) | 1
White blood cell count decreased (Investigations) | 1
White blood cell count increased (Investigations) | 1
Dehydration (Metabolism and nutrition disorders) | 1
Vitamin D deficiency (Metabolism and nutrition disorders) | 2
Muscle contracture (Musculoskeletal and connective tissue disorders) | 1
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1
Osteopenia (Musculoskeletal and connective tissue disorders) | 1
Fibroma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Clonus (Nervous system disorders) | 1
Tremor (Nervous system disorders) | 1
Agitation (Psychiatric disorders) | 1
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1
Aspiration (Respiratory, thoracic and mediastinal disorders) | 1
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 2
Bronchial secretion retention (Respiratory, thoracic and mediastinal disorders) | 1
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 1
Diaphragm muscle weakness (Respiratory, thoracic and mediastinal disorders) | 1
Diaphragmatic disorder (Respiratory, thoracic and mediastinal disorders) | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1
Increased bronchial secretion (Respiratory, thoracic and mediastinal disorders) | 1
Laryngeal stenosis (Respiratory, thoracic and mediastinal disorders) | 1
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 1
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 1
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 1
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 1
Tachypnoea (Respiratory, thoracic and mediastinal disorders) | 2
Wheezing (Respiratory, thoracic and mediastinal disorders) | 2
Dermatitis contact (Skin and subcutaneous tissue disorders) | 1
Dermatitis diaper (Skin and subcutaneous tissue disorders) | 3
Drug eruption (Skin and subcutaneous tissue disorders) | 1
Eczema (Skin and subcutaneous tissue disorders) | 1
Erythema (Skin and subcutaneous tissue disorders) | 2
Excessive granulation tissue (Skin and subcutaneous tissue disorders) | 2
Hair colour changes (Skin and subcutaneous tissue disorders) | 2
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1
Macule (Skin and subcutaneous tissue disorders) | 1
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 1
Papule (Skin and subcutaneous tissue disorders) | 1
Rash (Skin and subcutaneous tissue disorders) | 3
Rash erythematous (Skin and subcutaneous tissue disorders) | 1
Rash macular (Skin and subcutaneous tissue disorders) | 1
Rash papular (Skin and subcutaneous tissue disorders) | 1
Red man syndrome (Skin and subcutaneous tissue disorders) | 1
Skin exfoliation (Skin and subcutaneous tissue disorders) | 2
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 1
Skin hypopigmentation (Skin and subcutaneous tissue disorders) | 1
Skin irritation (Skin and subcutaneous tissue disorders) | 1
Skin ulcer (Skin and subcutaneous tissue disorders) | 1
Swelling face (Skin and subcutaneous tissue disorders) | 1
Gastrointestinal tube removal (Surgical and medical procedures) | 1
Post procedural drainage (Surgical and medical procedures) | 2
Flushing (Vascular disorders) | 1
Hypotension (Vascular disorders) | 1
Pallor (Vascular disorders) | 1
Vena cava thrombosis (Vascular disorders) | 1

LIMITATIONS AND CAVEATS:
Due to the small number of patients assessed in this study the results must be interpreted with caution.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
If no publication has occurred within 12 months of the completion of the study, the Investigator shall have the right to publish/present independently the results of the study. The Investigator shall provide the Sponsor with a copy of any such presentation/publication for comment at least 30 days before any presentation/submission for publication. If requested by the Sponsor, any presentation/submission shall be delayed up to 90 days, to allow the Sponsor to preserve its proprietary rights.